CLINICAL TRIAL: NCT07404358
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Dalargin for the Prevention of Postoperative Organ Dysfunction in Patients Undergoing High-Risk Abdominal Surgery
Brief Title: Dalargin for Prevention of Organ Disfunction in High-Risk Abdominal Surgery
Acronym: Dal-PROTECT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Botkin Hospital (Other)
Responsible Party: Principal Investigator, Anatolii Anatolievich Malyshev, Candidate og Medical Sciences, Head of the Department of Anesthesiology and Resuscitationa №62, role in study - principal Investigator, Botkin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BOTKIN-DAL-PROTECT-01; EC #6/25/5 (Other Grant/Funding Number: Independ Ethics Committee of the S.P. Botkin Moscow Multidisciplinary Sccientific and Clinical Center)
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Complications; Multiple Organ Failure; Abdominal Surgery
Keywords: Dalargin; Leu-enkephalin; Organ protection; Pharmacological preconditioning; Oxidative stress; Genetic polymorphis; High-risk surgery
MeSH Terms: conditions — Postoperative Complications; Multiple Organ Failure; Spinocerebellar ataxia 23 | interventions — enkephalin-Leu, Ala(2)-Arg(6)-; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a standart parallel-group, randomized, double-blind, placebo-controlled trial. Participants are allocated in a 1:1 ratio to either the experimental intervention (Dalargin) or the placebo control group. The study follows a fixed design without adaptive elements.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dalargin (Experimental): Patients in this arm receive a continuous intravenous of the study drug Dalargin (synthetic leucine-enkephalin analog) according to the predefined protocol
  Interventions: Drug: Dalargin
- Placebo (Placebo Comparator): Patients in this arm recive a continious intravenous infusion of 0.9% sodium chloride as a placebo, matching the volume and administration schedule of the active arm.
  Interventions: Other: 0.9 % NaCl

INTERVENTIONS:
Drug: Dalargin — Dalargin is a synthetic analog of the endogenous opioid peptide leucine-enkephalin. It is supplied as a lyophilized powder in vials containing 30 mg. For administration, the contents of one vial are reconstituted and diluted to a total volume of 300 ml with 0,9% sodium chloride (normal saline). The solution is administered as a continious intravenous infusion via an elastomeric infusion pump. The infusion starts after induction of anesthesia and continues for a total of 72 hours according to the following regimen: 8ml/hour (delivering 0.8 mg/hour) for the first 24 hours, followed by 4 ml/hour (delivering 0.4 mg/hour) for the subsequent 48 hours.
  Arms: Dalargin
Other: 0.9 % NaCl — A continious intravenous infusion of 0.9%sodium chloride used as a placebo control. It is prepared and administered in an identical manner (volume, duration, infusion device) as the active drug (Dalargin) to maintain blinding
  Other Names: Normal saline; Placebo; 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
Major abdominal surgeries (e.g., gastrectomy, pancreatectomy, colectomy) carry a high risk of life-threatening postoperative complications, including multiorgan disfunction syndrome (MODS), acute kidney injur (AKI), miocardial injury after non-cardiac surgery (MINS) and severe infections. These complications are driven by ischemia-reperfusion injury, leading to oxidative stress and a systemic inflammatory response. Despite advances in surgical and anesthetic techniques, there are no effective pharmacological strategies for personalized prevention of these events, which adversely affect recovery and survival.

In this context, opioid receptor agonist, particularly senthetic analogs of Leu-enkephalin such as Dalargin, have emerged as promising agents for pharmacologica preconditioning. Preclinical evidence suggests their ability to mitigate oxidative stress and inflammation by moduating key signaling pathways . The potential for these peptides to protect andothelial function and reduce organ damage presents a novel therapeutic avenue.

This study aims to clinically test the hypothesis that perioperative intravenous infusion of Dalargin reduce the incidence and severity of postoperative organ dysfunction. Patients undergoing high-risk abdominal surgery will be randomized to receive either a 72-hour continuous of Dalargin (following a defined dosage regimen) or an identical placebo infusion. the study will also integrate an assessment of genetic polymorphism ( e.g., in NRF2, OLR1, TLR9 genes) to explore personalized approaches to risk stratification and prevention.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled clinical trial. The study investigates the effects of a synthetic leucine-enkephalin analog (Dalargin) on oxidative distress, systemic inflammatory response, organ failure, and infectious complications in patients undergoing high-risk abdominal surgery (e.g. on the stomach, pancreas, or colon).

Objectives: The primary objective is to evaluate whether perioperative infusion of Dalargin reduces the incidence of a composite endpoint of postoperative organ dysfunction (including acute respiratory destress syndrome, acute kidney injury, and sepsis) . Secondary objectives include assessing its effects on biomarkers of oxidative stress (malondialdehyde, carbonylated proteins), inflammation (procalcitonin, interleukin-6, HMGB-1), and myocardial injury (high-sensitivity troponin T), as well asthe length of ICU and hospital stay.

Methods: A total of 200 patients aged 18-85 years (ASA I-III) scheduled for elective high-risk abdominal surgery ander general anesthesia will be randomized to recieve either Dalargin or placebo (0,9% sodium chloride). The study drug will be administered as a continious intravenous: 8 ml/hour for the first 24 hour, followed be 4 ml/hour for the next 48 hours, startinf after anesthesia induction. Patient outcomes will be evaluated using clinical scales (e.g., CPIS, KDIGO, APACHE II) and laboratory assessments. Additionally, genetic polymorphismis (NRF2, OLR1, TLR9, AGTR1, AQP1) will be analyzed to identify predictors of organ dysfunction and enable personalized risk stratification.

Scientific Navelty: This is the first study to comprehensively evaluate the organoprotective potential a synthetic enkephalin analog via pharmacological preconditioning in high-risk non-cardiac surgery, combining clinical endpoints with biomarker and genetic analysis to develop a personalized prevention strategy.

Sample Size Justification: The sample size of 200 participants (100/group) was calculated based on the anticipated incidence of the primary composite endpoint (postoperative organ dysfunction) in the control group. Based on previous similar studies and meta-analyses, we assume an event rate of 35% in the placebo group. We hypothesize that Dalargin will reduce this incidence to 20% (absolut risk reduction of 15%). With a two-sided alpha of 0.05 and 80% power, using a chisquared test, the required sample size is 178 participants. To account for a potential dropout rate of approximately 10%, the total sample size was increased to 200 partipitants. This sample size also provides adequate power (>80%) to detect clinically meaningful differences in key secondary endpoints, including the incidence of MINS (Myocardial Injury after non-cardiac Surgery) and changes in biomarker levels (e.g., interleukin-6)

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 85 years.
* Scheduled for elective high-risk abdominal surgery (e.g., gastrectome, pancreatectomy, colectomy) under general anesthesia.
* American Society of Anesthesiologists (ASA) physical status class I-III.
* Able to provide written informed consent.

Exclusion Criteria:

* ASA physical status class IV or V.
* Acute myocardial infarction within the past 6 month.
* Acute stroke within the past 6 month.
* Chronic heart failure NYHA class IV.
* Chronic kidney disease stage 3a or higher (according KDIGO)
* Active infectious disease.
* Any diagnosed phychiatric disorder (according ICD-10) confirmed be a psychiatrist.
* Any neuromuscular disease (according to ICD-10)
* Pregnancy or breastfeeding.
* Inability to undergo preoperative assessment.
* Previous enrollment in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Postoperative Complications | 7 days postoperatively
  Composite endpoin defined as the occurrence of at leats one of the follwing within the first 7 days after surgery: Miocardial injury after non-cardiac Surgery (MINS) (defined as an elevated high-sensitivity cardiac troponin T value with an ischemic feature, without requiring ischemic symptoms), Acute Kidney Injury (according to KDIGO criteria), Acute Respiratory Distress Syndrome (according to Berlin definition) or Sepsis (according to Sepsis - 3 criteria),

SECONDARY OUTCOMES:
Incident of acute respiratory distress syndrome (ARDS) | 7 days postoperatively
  Diagnosed according to the Berlin Definition (timing, origin, chest imaging, oxygenation)
Incidence of acute kidney injury (AKI) | 7 days postoperatively
  Defined and staged according to the kidney disease: improving Global Outcomes (KDIGO) criteris, based on serum creatinine and urine output.
Incident of sepsis | 7 days postoperatively
  Defined accorging to hte Sepsis-3 criteria as a life-threatening organ dysfunction caused by a dysregulated host response to infection
Plasma level of Interleukin-6 (IL-6) | 24 hours postoperatively
  Concentration measured in picograms per milliliter (pg/ml) using enzyme-linked immunosorbent assay (ELISA).
Plasma level of procalcitonin | 24 hours postoperatively
  Concentration measured in nanograms per milliliter (ng/ml)
Length of intensive care unit (ICU) stay | From surgery until ICU discharge, up to 30 days
  Total number of days spent in ICU from the day of surgery until discharge
Length of hospital stay | From surgery until hospital discharge, 30 days.
  Total numbers of days spent in the hospital from the day of surgery until discharge.
30-days all-cause mortality | 30 days postoperatively
  Death from any cause occurring within 30 days after the index surgery
Incidence of postoperative delirium | 7 days postoperatively
  Assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) or the 3-Minute Diagnostic Interview for (3D-CAM)
Level of oxidative stress marker (Malondialdehyde, MDA) | 2 days postoperatively
  Plasma concentration of malondialdehyde measured in micromoles per liter as a marker of lipid peroxidation
Chande in insulin resistance (HOMA-IR) | 5 days postoperatively
  Change in the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) index from baseline to the postoperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- S.P. Botkin Moscow Multidisciplinary Scientific and Clinical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No